CLINICAL TRIAL: NCT00277069
Title: INST: Phase I-II Study of Carboplatin, Vinorelbine and Capecitabine in Patients With Metastatic Breast Cancer
Brief Title: Phase I-II Study of Carboplatin, Vinorelbine and Capecitabine in Patients With Metastatic Breast Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of New Mexico (Other)
Responsible Party: Ian Rabinowitz, MD, University of New Mexico CRTC
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2899C
Record Dates: First submitted 2006-01-12; First posted 2006-01-13 (Estimated); Last update posted 2010-01-07 (Estimated); Status verified 2008-10

CONDITIONS: Breast; Cancer
Keywords: Breast metastatic
MeSH Terms: conditions — Neoplasms | interventions — Carboplatin; Vinorelbine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Carboplatin — Carboplatin given at 300mg/m2 IV over 30 minutes day 1, q 21 days
Device: Capecitabine — Capecitabine is administered at 1500mg/m2 PO qd in 2 divided doses day 1-14 q 21 days
  Other Names: Xeloda
Drug: Vinorelbine — Vinorelbine: 25mg/m2 IV over 10 minutes day 1, 8 q 21 days
  Other Names: Navelbine

SUMMARY:
1. Determine the response rate with this regimen in an anthracycline and taxane resistant cohort of patients.

DETAILED DESCRIPTION:
1. Determine the response rate with this regimen in an anthracycline and taxane resistant cohort of patients.
2. Determine a maximum tolerated dose of capecitabine in combination with vinorelbine and carboplatin for this patient population.
3. Determine the time to relapse after the administration of this regimen.

ELIGIBILITY:
Inclusion Criteria:

* Patient must have a histological diagnosis of breast cancer with metastasis.
* The metastatic disease should be confirmed by biopsy if clinically indicated.
* The patient must have measurable or evaluable disease.
* Age > 18 years and < 75 years.
* The patient may not have received prior therapy with vinorelbine, capecitabine, carboplatinum, or cisplatinum.
* The patient may have received herceptin previously.
* The patients must have previously received at least one cycle of chemotherapy.
* The patient must have received anthracycline and taxane containing chemotherapy in the past. This may be either in the adjuvant setting or for metastatic disease. Resistance is defined as progressive disease while on treatment, with or without an initial response, or relapse/progression within 6 months of completing chemotherapy.
* Performance status < 2.
* At least 3 weeks must have elapsed since the completion of prior radiation therapy, chemotherapy, or hormonal therapy. The patient must have recovered from all grade 3-4 associated toxicities at the time of registration. Measurable or evaluable disease must be outside the previous radiation field or a new lesion must be present.
* Patients must not receive concurrent hormonal, or biologic therapy, or radiation therapy to measurable or evaluable disease.
* The patient should not have uncontrolled CNS disease.
* Laboratory parameters: ANC > l500/ l, Platelets >100 000/ l, creatinine < 2.0, bilirubin < 2.0
* Informed consent.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2000-05; Primary Completion 2005-03 (Actual); Study Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
Measurable disease: Bidimensionally measurable lesions with clearly defined margins by 1) palpation with both diameters greater than 1 cm, 2) CT, MRI with both diameters greater than the distance between cuts of the imaging study. | disease progression or unacceptable toxicities

CONTACTS AND LOCATIONS:
Overall Officials: Ian Rabinowitz, MD, Principal Investigator — University of New Mexico
Locations (1):
- University of New Mexico, Albuquerque, New Mexico, United States